CLINICAL TRIAL: NCT05825859
Title: Total Body Perfusion in Patients With Chest Pain
Acronym: KOVERI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Juhani Knuuti, Professor, Turku University Hospital
Other Study IDs: KOVERI
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Purpose of this study is to better understand changes in obstructive coronary artery disease in different organs other than the heart such as the brain and the kidneys using a new generation total body PET scanner.

DETAILED DESCRIPTION:
Patients with chest pain and suspected CAD will be studied using total body PET imaging with O15-water perfusion imaging

ELIGIBILITY:
Inclusion Criteria:

* Documented history of chest pain with CT imaging showing a potential for obstructive coronary artery disease
* Ability to sustain adenosine injection 0.14 mg/kg/min

Exclusion Criteria:

* Second or third degree AV-block without pacemaker
* Sick sinus syndrome
* Consumption of coffee or aminophylline within 12 hours of administration
* Recent use of dipyridmole or dipyridamole-containing medications
* Known hypersensitivity to adenosine
* Unstable acute MI or acute coronary artery syndrome, and prior cardiac transplantation
* Active wheezing and bronchospasm
* Sinus bradycardia with HR<40 bmp

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Finnish people that have history of chest pain and for which there have been done CTA which shows a possibility for obstructive coronary artery disease. All people in the study population have came to a diagnostic radiowater imgaing to know if there is significant obsturction of the coronary arteries.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Perfusion in heart, brain and kidneys during rest and adenosine stress, and their associations with psychologic factors and anginal symptoms | The imaging day
  Multiorgan perfusion changes in patients with chest pain

SECONDARY OUTCOMES:
The association between perfusion in heart, brain and kidneys, and adverse events during five year follow-up | Five year follow-up after the imaging
  Multiorgan perfusion changes in patients with chest pain as related to outcome

CONTACTS AND LOCATIONS:
Overall Officials: Juhani Knuuti, MD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No